CLINICAL TRIAL: NCT01746186
Title: The Energy Balance Study
Status: Completed | Type: Observational
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Sarah Schumacher, Director, University of South Carolina
Other Study IDs: Pro00009704
Record Dates: First submitted 2012-11-26; First posted 2012-12-10 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Total Energy Expenditure,Total Energy Intake

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 21-35 years of age: 200 Men and 200 women: Ages 21-27 and Ages 28-35, BMI: 20-35,living in the Columbia, SC area.

SUMMARY:
The purpose of this study if to determine the specific contributions of energy intake and energy expenditure to changes in body weight and fat.

DETAILED DESCRIPTION:
1. Changes in body weight and fat will be positively associated with increases in total energy intake.
2. Changes in body weight and fat will be positively associated with decreases in total energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 20-35 *Note : For participants that come to Orientation, we are allowing participants with a variance of 0.1 either way in the BMI range: 19.9 - 35.1

  * 21-35 years of age
  * Men and women
  * Email address
  * Access to a phone

Exclusion Criteria:

* Currently on medications to lose weight

  * >90th percentile on the Brief Symptom Inventory (BSI)
  * Planning to move from the Greater Columbia area in the next 15 months
  * Other medical, psychiatric or behavioral factors that in the judgment of the principal investigator may interfere with study participation or the ability to follow the intervention protocol.
  * Changed birth control status in past 3 months
  * Currently taking birth control but plan to stop taking it within the next 12 months or are planning to start taking birth control in the next 12 months
  * Planning to have weight loss surgery
  * Started or stopped smoking in the past 6 months
  * Blood pressure ≥ 150/90
  * Blood glucose ≥ 145 mg/dL @ orientation
  * Blood glucose ≥ 126 mg/dL @ B3
  * Total cholesterol ≥ 240 mg/dl with LDL-C ≥ 190 mg/dl or Triglyceride levels ≥ 300 mg/dL
  * Currently diagnosed with or taking medications for a major chronic health condition
  * Presence of an eating disorder
  * Currently participating in another study

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 400 participants will take part in the Energy Balance Study; 200 men and 200 women from 2 age groups: Ages 21-27 and Ages 28-35. A subsample of 200 will be randomized for doubly labeled water recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
variation in total energy expenditure and variation in total energy intake contribute to changes in body weight and fat among young adults | two years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Blair, Ph.D, Principal Investigator — University of South Carolina; Greg Hand, Ph.D, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Meyer JD, Ellingson LD, Buman MP, Shook RP, Hand GA, Blair SN. Current and 1-Year Psychological and Physical Effects of Replacing Sedentary Time With Time in Other Behaviors. Am J Prev Med. 2020 Jul;59(1):12-20. doi: 10.1016/j.amepre.2020.02.018. Epub 2020 May 14. PMID 32418803
- [Derived] Shook RP, Hand GA, Drenowatz C, Hebert JR, Paluch AE, Blundell JE, Hill JO, Katzmarzyk PT, Church TS, Blair SN. Low levels of physical activity are associated with dysregulation of energy intake and fat mass gain over 1 year. Am J Clin Nutr. 2015 Dec;102(6):1332-8. doi: 10.3945/ajcn.115.115360. Epub 2015 Nov 11. PMID 26561620
- [Derived] Shook RP, Gribben NC, Hand GA, Paluch AE, Welk GJ, Jakicic JM, Hutto B, Burgess S, Blair SN. Subjective Estimation of Physical Activity Using the International Physical Activity Questionnaire Varies by Fitness Level. J Phys Act Health. 2016 Jan;13(1):79-86. doi: 10.1123/jpah.2014-0543. Epub 2015 Apr 21. PMID 25898394
- [Derived] Shook RP, Hand GA, Paluch AE, Wang X, Moran R, Hebert JR, Lavie CJ, Blair SN. Moderate cardiorespiratory fitness is positively associated with resting metabolic rate in young adults. Mayo Clin Proc. 2014 Jun;89(6):763-71. doi: 10.1016/j.mayocp.2013.12.017. Epub 2014 May 5. PMID 24809761